CLINICAL TRIAL: NCT02364206
Title: Phase I/II Study of LY2228820 With Radiotherapy Plus Concomitant TMZ in the Treatment of Newly Diagnosed Glioblastoma
Brief Title: Study of LY2228820 With Radiotherapy Plus Concomitant TMZ in the Treatment of Newly Diagnosed Glioblastoma
Acronym: GLYRad
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: National Cancer Institute, France (Other Government); ARC Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-005442-11
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Adult Glioblastoma
Keywords: newly diagnosed glioblastoma; p38 MAPK inhibitor; temozolomide; radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — ralimetinib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2228820 + TMZ + Radiotherapy (Experimental): addition of LY2228820 to standard radiotherapy and concomitant treatment by temozolomide (TMZ).
  LY2228820 will be administered orally for two 28 day cycles, from one week before the beginning of radiotherapy, and during standard chemoradiotherapy. Three dose levels of LY2228820 will be tested.
  After a 4 week break after concomitant treatment, patient were then received up to 6 cycles of adjuvant TMZ according to the standard 5-day schedule every 28 days .
  Interventions: Drug: LY2228820; Drug: Temozolomide; Radiation: radiotherapy

INTERVENTIONS:
Drug: LY2228820
  Other Names: ralimetinib
Drug: Temozolomide
  Other Names: TMZ
Radiation: radiotherapy

SUMMARY:
Glioblastomas are extremely resistant to treatment, including radiotherapy and/or chemotherapy. Mitogen-activated protein kinase (MAPK) cascades are key signaling pathways involved in the regulation of normal cell proliferation, survival and differentiation. Activation of p38 MAPK has been associated with a poor prognosis among patients with glioblastoma during the temozolomide (TMZ) era and represents a compensatory response by tumor cell to environmental stress such as radiation or chemotherapy.

LY2228820 is a potent and selective inhibitor of p38 MAPK, and reduces phosphorylation of its cellular target, MAPK-activated protein kinase 2 (MAPKAPK-2) . LY2228820 is a good candidate to target malignant glioma resistance to the gold standard treatment combining radiation and TMZ by acting on both tumor and stromal cells.

The primary objectives of this study were to determine the recommended dose of LY2228820 in combination with TMZ and radiotherapy during chemoradiotherapy period (phase I) and to estimate the 6-month progression free survival (PFS) rate of patients treated with LY2228820 when administered at the recommended dose in combination with radiotherapy and concomitant TMZ (phase II)

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and histologically confirmed glioblastoma
* Recursive partitioning analysis (RPA) class III or IV
* Age > or = 18 years and < 75 years of age
* Life expectancy > or = 6 months
* Patient must have at least 1 formalin fixed paraffin embedded tumor tissue block representative of glioblastoma available for pathology central review and biomarker exploration
* Adequate hematologic (absolute neutrophil count (ANC) > or = 1.5 x 109/L, platelet count > or = 100 x 109/L, hemoglobin > or = 10 g/dL ), renal (creatinine > or = 1.25 x ULN ), and hepatic function (total bilirubin < or = 1.5 x ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < or = 2.5 x ULN)
* Patients who were receiving corticosteroids had to receive a stable or decreasing dose for at least 14 days before enrollment
* Patients must be able to swallow and retain oral medication
* Women must have a negative serum pregnancy test less than 7 days prior to the first dose of study drug
* Both men and women of reproductive potential agree to use approved contraception during the study and for 6 months after discontinuation of study treatment.
* Willing and able to comply with the protocol as judged by the investigator
* Patients must provide written consent

Exclusion Criteria:

* Any prior chemotherapy (including carmustine-containing wafers) or immunotherapy (including vaccine therapy )
* Any prior radiotherapy to the brain
* Any contraindication to temozolomide listed in the local label
* Have had, in the judgment of the investigator, a major bowel resection that would alter oral drug absorption
* Have a diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Have previously completed or withdrawn from this study or any other study investigating LY2228820
* Are receiving, in the judgment of the investigator, concurrent administration of immunosuppressive therapy
* Diarrhea of any cause CTCAE > or = grade 2
* Current or recent (within 30 days of enrollment) treatment with another investigational drug or participation in another investigational study
* History of other malignancy within 5 years prior enrollment except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Pregnant or nursing (lactating) woman, or fertile women unwilling or unable to use effective means of contraception
* Psychiatric illness / social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance / pill diary

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) (phase I) of LY2228820 in combination with TMZ and radiotherapy during chemoradiotherapy period | from D1 Week 0 (first dose of LY2228820) to D63 Week 8.
  defined as the highest dose tested in which a dose limiting toxicity (DLT) is experienced by no more than 33% of patients during chemoradiotherapy period.
6-month Progression Free Survival (PFS) rate (phase II) defined as the rate of patients who not presented a progression at 6 months from the first dose of LY2228820 | 6 months from the first dose of LY2228820

SECONDARY OUTCOMES:
Safety profile according to NCI Common Toxicity Criteria for Adverse Effect (CTCAE) criteria version 4.03. | from baseline to 30 days after treatment (concomitant and adjuvant treatment) (week 35)
PFS | from the first dose of LY2228820 to disease progression or death for any reason, up to 24 months
  disease progression assessed per Response Assessment in Neuro-Oncology (RANO) criteria
Overall Survival | from the first dose of LY2228820 to death, up to 24 months
12-month PFS rate defined as the rate of patients who not presented a progression at 12 months from the first dose of LY2228820 | 12 months from the first dose of LY2228820
Objective response rate according to RANO criteria for patients with incomplete resection or only biopsy | from the first dose of LY2228820 to treatment completion
The neurologic status evaluated by clinical assessment and Mini-Mental State Examination (MMSE) and evaluation of corticosteroid dosage | from baseline to progression, up to 24 months
Pharmacokinetic of LY2228820 and TMZ (AUC0-12h) | D7 Week 0, D28 Week 3, D35 Week 4
MAPKAPK-2 activation | baseline (tumor) D1 D7 week 0, D28 Week 3, D35 Week 4 (PBMCs)
  in tumor and stromal cells and Peripheral Blood Mononucleated Cells (PBMCs)
Validated biomarker of glioblastoma (MGMT, IDH1 (isocitrate dehydrogenase 1), pTEN (phosphatase and tensin homolog), p53) | baseline
  on tumor

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Pr, Principal Investigator — Centre Jean Perrin
Locations (6):
- France (6):
  - CHU Amiens Sud-Salouel, Amiens
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Paul Strauss, Strasbourg